CLINICAL TRIAL: NCT02437136
Title: A Phase 1b/2, Open-label, Dose Escalation Study of Entinostat in Combination With Pembrolizumab in Patients With Non-small Cell Lung Cancer, With Expansion Cohorts in Patients With Non-small Cell Lung Cancer, Melanoma, and Mismatch Repair-Proficient Colorectal Cancer
Brief Title: Ph1b/2 Dose-Escalation Study of Entinostat With Pembrolizumab in Non-small Cell Lung Cancer (NSCLC) With Expansion Cohorts in NSCLC, Melanoma, and Colorectal Cancer (CRC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Syndax Pharmaceuticals (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNDX-275-0601; KN 142 (Other: Merck & Co.)
Record Dates: First submitted 2015-04-27; First posted 2015-05-07 (Estimated); Results first posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Non-Small Cell Lung Cancer; Melanoma; Mismatch Repair-Proficient Colorectal Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Melanoma | interventions — entinostat; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Phase 1b (Dose Escalation): Entinostat 3 mg Weekly + Pembrolizumab (Experimental): Participants with NSCLC will receive entinostat 3 mg administered orally weekly (Days 1, 8, and 15 of each 21-day cycle) along with pembrolizumab 200 mg via intravenous (IV) infusion once every 3 weeks (Day 1 of each 21-day cycle).
  Interventions: Drug: entinostat; Drug: pembrolizumab
- Phase 1b (Dose Escalation): Entinostat 5 mg Weekly + Pembrolizumab (Experimental): Participants with NSCLC will receive entinostat 5 mg administered orally weekly (Days 1, 8, and 15 of each 21-day cycle) along with pembrolizumab 200 mg via IV infusion once every 3 weeks (Day 1 of each 21-day cycle).
  Interventions: Drug: entinostat; Drug: pembrolizumab
- Phase 1b (Dose Confirmation): Entinostat 5 mg Weekly + Pembrolizumab (Experimental): Participants with NSCLC will receive entinostat 5 mg administered orally weekly (Days 1, 8, and 15 of each 21-day cycle) along with pembrolizumab 200 mg via IV infusion once every 3 weeks (Day 1 of each 21-day cycle).
  Interventions: Drug: entinostat; Drug: pembrolizumab
- Phase 2, Cohort 1: Entinostat 5 mg Weekly + Pembrolizumab (Experimental): Participants with NSCLC with squamous cell or adenocarcinoma histology who had not been treated with a programmed cell death receptor-1 (PD-1)- or programmed cell death ligand-1 (PD-L1)-blocking antibody, will receive entinostat 5 mg administered orally weekly (Days 1, 8, and 15 of each 21-day cycle) along with pembrolizumab 200 mg via IV infusion once every 3 weeks (Day 1 of each 21-day cycle).
  Interventions: Drug: entinostat; Drug: pembrolizumab
- Phase 2, Cohort 2: Entinostat 5 mg Weekly + Pembrolizumab (Experimental): Participants with NSCLC (any histology) who has previously been treated with and unequivocally progressed on either a PD-1- or PD-L1-blocking antibody, will receive entinostat 5 mg administered orally weekly (Days 1, 8, and 15 of each 21-day cycle) along with pembrolizumab 200 mg via IV infusion once every 3 weeks (Day 1 of each 21-day cycle).
  Interventions: Drug: entinostat; Drug: pembrolizumab
- Phase 2, Cohort 3: Entinostat 5 mg Weekly + Pembrolizumab (Experimental): Participants with melanoma who has previously been treated with and unequivocally progressed on either a PD-1- or PD-L1-blocking antibody, will receive entinostat 5 mg administered orally weekly (Days 1, 8, and 15 of each 21-day cycle) along with pembrolizumab 200 mg via IV infusion once every 3 weeks (Day 1 of each 21-day cycle).
  Interventions: Drug: entinostat; Drug: pembrolizumab
- Phase 2, Cohort 4: Entinostat 5 mg Weekly + Pembrolizumab (Experimental): Participants with CRC (mismatch repair-proficient) who had not been previously treated with a PD-1- or PD-L1-blocking antibody, received entinostat 5 mg administered orally weekly (Days 1, 8, and 15 of each 21-day cycle) along with pembrolizumab 200 mg via IV infusion once every 3 weeks (Day 1 of each 21-day cycle).
  Interventions: Drug: entinostat; Drug: pembrolizumab

INTERVENTIONS:
Drug: entinostat — An orally available histone deacetylases inhibitor (HDACs)
  Other Names: SNDX-275; MS-275
Drug: pembrolizumab — A selective humanized monoclonal antibody (mAb)
  Other Names: Keytruda; MK-3475; SCH 900475

SUMMARY:
The purpose of this study is to determine the safety and tolerability of entinostat used in combination with pembrolizumab in participants with NSCLC. Additionally, the purpose of the study is to assess how effective entinostat and pembrolizumab are in combination in participants with NSCLC, Melanoma, and Mismatch-Repair Proficient CRC.

ELIGIBILITY:
Inclusion Criteria:

Participants with NSCLC:

1. Has histologically- or pathologically-confirmed recurrent/metastatic NSCLC.
2. If has adenocarcinoma, required to have previously been tested for anaplastic lymphoma kinase (ALK) rearrangements and epidermal growth factor receptor (EGFR) mutations, with results available for collection in this study, and, if positive, has been treated with prior epidermal growth factor receptor (EGFR) or ALK therapy.
3. Received at least 1 chemotherapeutic regimen in the advanced/metastatic setting and experienced documented, unequivocal progressive disease by either RECIST 1.1 or clinical assessment. Additional requirements related to prior treatments applied and may have been dependent on mutational status.
4. Participants with NSCLC enrolled in Cohort 1 of the Expansion Phase should not have been previously treated with a PD-1/PD-L1-blocking antibody.

   Participants in Expansion Phase, Cohorts 2 (NSCLC) and 3 (Melanoma):
5. Previously treated with a PD-1/PD-L1-blocking antibody and experienced documented, unequivocal radiographic progression of disease by irRECIST, or similar criteria during or within 12 weeks after last dose of such treatment. Participants must have received at least 6 weeks of PD-1/PD-L1 therapy for Cohort 2 and at least 8 weeks of PD-1/PD-L1 therapy for Cohort 3.

   Participants with Melanoma:
6. In addition to having been previously treated with a PD-1/PD-L1-blocking antibody, has a histologically- or cytologically-confirmed diagnosis of unresectable or metastatic melanoma and experienced unequivocal progressive disease during treatment with a Serine/threonine-protein kinase B-Raf (BRAF) inhibitor if BRAF V600 mutation-positive. Treatment with BRAF inhibitor may occur after treatment with the checkpoint inhibitor.

   Participants in Expansion Phase, Cohort 4 (CRC):
7. Received at least 1 chemotherapeutic regimen in the advanced/metastatic setting and experienced documented, unequivocal progressive disease by either RECIST 1.1 or clinical assessment. Must have documented mismatch repair-proficient colon cancer as determined by either immunohistochemistry for mismatch repair proteins or polymerase chain reaction (PCR)-based functional microsatellite instability. Participants with CRC enrolled in Cohort 4 should not have been previously treated with a PD-1/PD-L1-blocking antibody (that is, pembrolizumab, nivolumab, MEDI4736, or GNE PDL1 [MPDL3280A]).

   All Participants:
8. Aged 18 years or older on the day written informed consent is given.
9. If has brain metastases, must have stable neurologic status following local therapy for at least 4 weeks without the use of steroids or on stable or decreasing dose of ≤10 milligrams (mg) daily prednisone (or equivalent), and must be without neurologic dysfunction that would confound the evaluation of neurologic and other AEs.
10. Evidence of locally recurrent or metastatic disease based on imaging studies within 28 days before the first study drug dose:

    * At least 1 measurable lesion ≥20 mm by conventional techniques or ≥10 mm by spiral computed tomography (CT) scan or magnetic resonance imaging (MRI), with the last imaging performed within 28 days before the first study drug dose. If there is only 1 measurable lesion and it is located in previously irradiated field, it must have demonstrated unequivocal progression according to RECIST, version 1.1.
11. If receiving radiation therapy, has a 2-week washout period following completion of the treatment prior to receiving the first study drug dose and continues to have at least 1 measurable lesion, per above criterion.
12. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
13. Has acceptable renal and hepatic function and stable hematologic and coagulation status.
14. Female participants must not be pregnant. If a participants is of childbearing potential, the participant must agree to use effective contraception, as defined in the protocol, during the study and for 120 days after the last dose of study drug.
15. If male, agrees to use an adequate method of contraception starting from the first dose of study drug through 120 days after the last dose of study drug.
16. Experienced resolution of toxic effect(s) of the most recent prior chemotherapy to Grade 1 or less (except alopecia). If participant underwent major surgery or radiation therapy of >30 gray (Gy), they must have recovered from the toxicity and/or complications from the intervention.
17. Willing to have fresh tumor samples collected during screening and at other time points designated as mandatory, per the Schedule of Study Assessments.
18. Able to understand and give written informed consent and comply with study procedures.

Exclusion Criteria:

Participants meeting any of the following criteria are not eligible for study participation:

1. Diagnosis of immunodeficiency or receiving systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug. The use of physiologic doses of corticosteroids may be approved after consultation with the Sponsor.
2. Active autoimmune disease that has required systemic treatment in past 2 years (that is, with disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (for example, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.
3. History of interstitial lung disease (ILD).
4. Allergy to benzamide or inactive components of entinostat.
5. History of allergies to any active or inactive ingredients of pembrolizumab or severe hypersensitivity (≥Grade 3) to pembrolizumab.
6. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator, including, but not limited to:

   * Myocardial infarction or arterial thromboembolic events within 6 months prior to baseline or severe or unstable angina, New York Heart Association (NYHA) Class III or IV disease, or a QTc interval > 470 milliseconds (msec).
   * Uncontrolled heart failure or hypertension, uncontrolled diabetes mellitus, or uncontrolled systemic infection.
   * Another known additional malignancy that is progressing or requires active treatment (excluding adequately treated basal cell carcinoma, squamous cell of the skin, cervical intraepithelial neoplasia [CIN]/cervical carcinoma in situ or melanoma in situ, or ductal carinoma in situ of the breast). Prior history of other cancer is allowed, as long as there is no active disease within the prior 5 years.
   * Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
   * Active infection requiring systemic therapy.
   * Known active central nervous system (CNS) metastases and/or carcinomatous meningitis.

   Note: Participants with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging [using the identical imaging modality for each assessment, either MRI or CT scan] for at least 4 weeks prior to the first dose of study drug and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 2 weeks prior to the first dose of study drug or are on stable or decreasing dose of ≤10 mg daily prednisone (or equivalent). This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
7. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
8. Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
9. Received a live virus vaccination within 30 days of the first dose of treatment.
10. Prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to baseline or who has not recovered (that is, ≤Grade 1 or at baseline) from AEs due to agents administered more than 4 weeks earlier.
11. Prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study baseline or who has not recovered (that is, ≤Grade 1 or at baseline) from AEs due to a previously administered agent.

    Note: Participants with ≤Grade 2 neuropathy or ≤Grade 2 alopecia are an exception to this criterion and may qualify for the study.

    Note: If participant underwent major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
12. Received transfusion of blood products (including platelets or red blood cells) or administration of colony stimulating factors (including granulocyte-colony stimulating factor [G-CSF], granulocyte macrophage-colony stimulating factor [GM-CSF], or recombinant erythropoietin) within 4 weeks prior to the first dose of study drug.
13. Currently receiving treatment with any other agent listed on the prohibited medication list such as valproic acid, or other systemic cancer agents within 14 days of the first dose of treatment.
14. If female, is pregnant, breastfeeding, or expecting to conceive, or if male, expect to father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study drug.
15. Known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies).
16. Known active hepatitis B (for example, hepatitis B surface antigen-reactive) or hepatitis C (for example, hepatitis C virus ribonucleic acid [qualitative]).
17. For CRC expansion cohort, no prior history of malignant bowel obstruction requiring hospitalization in the 6 months prior to enrollment
18. For the CRC expansion cohort, history of uncontrolled ascites, defined as symptomatic ascites and/or repeated paracenteses for symptom control in the past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2015-08-26 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2022-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pasi A Janne, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (11):
- United States (11):
  - Yale University, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - University of Maryland, Marlene and Stewart Greenbaum Cancer Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Dana Farber Cancer Institution, Boston, Massachusetts
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - St Luke's University Health Network, Easton, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee

REFERENCES:
- [Background] Simon R. Optimal two-stage designs for phase II clinical trials. Control Clin Trials. 1989 Mar;10(1):1-10. doi: 10.1016/0197-2456(89)90015-9. PMID 2702835
- [Derived] Hellmann MD, Janne PA, Opyrchal M, Hafez N, Raez LE, Gabrilovich DI, Wang F, Trepel JB, Lee MJ, Yuno A, Lee S, Brouwer S, Sankoh S, Wang L, Tamang D, Schmidt EV, Meyers ML, Ramalingam SS, Shum E, Ordentlich P. Entinostat plus Pembrolizumab in Patients with Metastatic NSCLC Previously Treated with Anti-PD-(L)1 Therapy. Clin Cancer Res. 2021 Feb 15;27(4):1019-1028. doi: 10.1158/1078-0432.CCR-20-3305. Epub 2020 Nov 17. PMID 33203644
- See also: CTCAE v. 4.03 — http://www.hrc.govt.nz/sites/default/files/CTCAE%20manual%20-%20DMCC.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 2 phases, a Dose Escalation/Confirmation Phase (Phase 1b) and an Expansion Phase (Phase 2).
Pre-assignment Details: Per protocol, 9 participants in the Confirmation Phase who rolled over to Cohort 2, and the other 7 participants who rolled over to Cohort 1 in the Expansion Phase, were counted in the Expansion Phase Population rather than in the Escalation/Confirmation Phase Population for the purpose of collecting data.
Groups:
- Phase 1b (Dose Escalation): Entinostat 3 mg Weekly + Pembrolizumab: Participants with non-small cell lung cancer (NSCLC) received entinostat 3 milligrams (mg) administered orally weekly (Days 1, 8, and 15 of each 21-day cycle) along with pembrolizumab 200 mg via intravenous (IV) infusion once every 3 weeks (Day 1 of each 21-day cycle).
- Phase 1b (Dose Escalation): Entinostat 5 mg Weekly + Pembrolizumab; Phase 1b (Dose Confirmation): Entinostat 5 mg Weekly + Pembrolizumab: Participants with NSCLC received entinostat 5 mg administered orally weekly (Days 1, 8, and 15 of each 21-day cycle) along with pembrolizumab 200 mg via IV infusion once every 3 weeks (Day 1 of each 21-day cycle).
- Phase 2, Cohort 1: Entinostat 5 mg Weekly + Pembrolizumab: Participants with NSCLC with squamous cell or adenocarcinoma histology who had not been treated with a programmed cell death receptor-1 (PD-1)- or programmed cell death ligand-1 (PD-L1)-blocking antibody, received entinostat 5 mg administered orally weekly (Days 1, 8, and 15 of each 21-day cycle) along with pembrolizumab 200 mg via IV infusion once every 3 weeks (Day 1 of each 21-day cycle).
- Phase 2, Cohort 2: Entinostat 5 mg Weekly + Pembrolizumab: Participants with NSCLC (any histology) who had previously been treated with and unequivocally progressed on either a PD-1- or PD-L1-blocking antibody, received entinostat 5 mg administered orally weekly (Days 1, 8, and 15 of each 21-day cycle) along with pembrolizumab 200 mg via IV infusion once every 3 weeks (Day 1 of each 21-day cycle).
- Phase 2, Cohort 3: Entinostat 5 mg Weekly + Pembrolizumab: Participants with melanoma who had previously been treated with and unequivocally progressed on either a PD-1- or PD-L1-blocking antibody, received entinostat 5 mg administered orally weekly (Days 1, 8, and 15 of each 21-day cycle) along with pembrolizumab 200 mg via IV infusion once every 3 weeks (Day 1 of each 21-day cycle).
- Phase 2, Cohort 4: Entinostat 5 mg Weekly + Pembrolizumab: Participants with colorectal cancer (CRC) (mismatch repair-proficient) who had not been previously treated with a PD-1- or PD-L1-blocking antibody, received entinostat 5 mg administered orally weekly (Days 1, 8, and 15 of each 21-day cycle) along with pembrolizumab 200 mg via IV infusion once every 3 weeks (Day 1 of each 21-day cycle).
Period: Dose Escalation/Confirmation (Phase 1b)
Arm/Group | Phase 1b (Dose Escalation): Entinostat 3 mg Weekly + Pembrolizumab | Phase 1b (Dose Escalation): Entinostat 5 mg Weekly + Pembrolizumab | Phase 1b (Dose Confirmation): Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 1: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 2: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 3: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 4: Entinostat 5 mg Weekly + Pembrolizumab
Started | 6 | 7 | 9 | 0 | 0 | 0 | 0
Received at Least 1 Dose of Study Drug | 6 | 7 | 9 | 0 | 0 | 0 | 0
Completed | 2 | 7 (Rolled over to 'Phase 2, Cohort 1: Entinostat 5 mg Weekly + Pembrolizumab') | 9 (Rolled over to 'Phase 2, Cohort 2: Entinostat 5 mg Weekly + Pembrolizumab') | 0 | 0 | 0 | 0
Not Completed | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 4 | 0 | 0 | 0 | 0 | 0 | 0
Period: Expansion (Phase 2)
Arm/Group | Phase 1b (Dose Escalation): Entinostat 3 mg Weekly + Pembrolizumab | Phase 1b (Dose Escalation): Entinostat 5 mg Weekly + Pembrolizumab | Phase 1b (Dose Confirmation): Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 1: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 2: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 3: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 4: Entinostat 5 mg Weekly + Pembrolizumab
Started | 0 | 0 | 0 | 18 (7 participants rolled over from 'Phase 1b (Dose Escalation): Entinostat 5 mg Weekly + Pembrolizumab'.) | 76 (9 participants rolled over from 'Phase 1b (Dose Confirmation): Entinostat 5 mg Weekly + Pembrolizumab'.) | 53 | 38
Received at Least 1 Dose of Study Drug | 0 | 0 | 0 | 18 | 76 | 53 | 38
Completed | 0 | 0 | 0 | 5 | 11 | 17 | 10
Not Completed | 0 | 0 | 0 | 13 | 65 | 36 | 28
Not completed — Death | 0 | 0 | 0 | 6 | 37 | 29 | 24
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 7 | 25 | 4 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 3 | 3 | 2

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of either study drug, entinostat, or pembrolizumab.
Groups:
- Phase 1b (Dose Escalation): Entinostat 3 mg Weekly + Pembrolizumab: Participants with NSCLC received entinostat 3 mg administered orally weekly (Days 1, 8, and 15 of each 21-day cycle) along with pembrolizumab 200 mg via IV infusion once every 3 weeks (Day 1 of each 21-day cycle).
- Phase 2, Cohort 1: Entinostat 5 mg Weekly + Pembrolizumab: Participants with NSCLC with squamous cell or adenocarcinoma histology who had not been treated with a PD-1- or PD-L1-blocking antibody, received entinostat 5 mg administered orally weekly (Days 1, 8, and 15 of each 21-day cycle) along with pembrolizumab 200 mg via IV infusion once every 3 weeks (Day 1 of each 21-day cycle).
- Total: Total of all reporting groups
Arm/Group | Phase 1b (Dose Escalation): Entinostat 3 mg Weekly + Pembrolizumab | Phase 2, Cohort 1: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 2: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 3: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 4: Entinostat 5 mg Weekly + Pembrolizumab | Total
Number analyzed (Participants) | 6 | 18 | 76 | 53 | 38 | 191
Age, Customized [Count of Participants; unit: Participants]
  Age: 44 years and younger | 0 | 1 | 1 | 6 | 6 | 14
  Age: 45 to 64 years | 1 | 7 | 35 | 23 | 24 | 90
  Age: 65 to 74 years | 5 | 7 | 25 | 14 | 6 | 57
  Age: 75 years and older | 0 | 3 | 15 | 10 | 2 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 8 | 36 | 21 | 14 | 80
  Male | 5 | 10 | 40 | 32 | 24 | 111
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 2 | 1 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 3 | 3 | 5 | 12
  White | 4 | 15 | 66 | 47 | 32 | 164
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 5 | 2 | 1 | 10

OUTCOME MEASURES:

1. Primary Outcome: Phase 2: Objective Response Rate (ORR), as Assessed Using Immune Response RECIST (irRECIST)
Description: The ORR was defined as the percentage of participants with confirmed complete response (CR) or partial response (PR). CR: Complete disappearance of all lesions (whether measurable or not) and no new lesions. All measurable lymph nodes also must have a reduction in short axis to <10 millimeters (mm). PR: Sum of the diameters (longest for non-nodal lesions, shortest for nodal lesions) of target and new measurable lesions decreases ≥30%. For purposes of analysis, 1 month was considered to be 30.4375 days.
Time Frame: From date of randomization to date of progression (up to 765 days)
Population: Full analysis set (FAS) included all enrolled participants excluding those that did not receive at least 1 dose of entinostat and pembrolizumab or lacked baseline data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2, Cohort 1: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 2: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 3: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 4: Entinostat 5 mg Weekly + Pembrolizumab
Number analyzed (Participants) | 18 | 76 | 53 | 37
percentage of participants | 22.2 [6.4 to 47.6] | 9.2 [3.8 to 18.1] | 18.9 [9.4 to 32.0] | 5.4 [0.7 to 18.2]

2. Secondary Outcome: Phase 2: Clinical Benefit Rate (CBR), as Assessed Using irRECIST
Description: The CBR was defined as the percentage of participants with a confirmed CR, PR, or stable disease (SD) lasting for at least 6 months. CR: Complete disappearance of all lesions (whether measurable or not) and no new lesions. All measurable lymph nodes also must have a reduction in short axis to <10 mm. PR: Sum of the diameters (longest for non-nodal lesions, shortest for nodal lesions) of target and new measurable lesions decreases ≥30%. SD: Sum of the diameters (longest for nonnodal lesions, shortest for nodal lesions) of target and new measurable lesions neither CR, PR, (compared to baseline) or progressive disease (PD) (compared to nadir).
Time Frame: 6 months
Population: FAS included all enrolled participants excluding those that did not receive at least 1 dose of entinostat and pembrolizumab or lacked baseline data. Data were not censored for CBR analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase 2, Cohort 4: Entinostat 5 mg Weekly + Pembrolizumab: Participants with CRC (mismatch repair-proficient) who had not been previously treated with a PD-1- or PD-L1-blocking antibody, received entinostat 500 mg administered orally weekly (Days 1, 8, and 15 of each 21-day cycle) along with pembrolizumab 200 mg via IV infusion once every 3 weeks (Day 1 of each 21-day cycle).
Arm/Group | Phase 2, Cohort 1: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 2: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 3: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 4: Entinostat 5 mg Weekly + Pembrolizumab
Number analyzed (Participants) | 18 | 76 | 53 | 37
percentage of participants | 33.3 [13.3 to 59.0] | 14.5 [7.5 to 24.4] | 35.8 [23.1 to 50.2] | 8.1 [1.7 to 21.9]

3. Secondary Outcome: Phase 2: CBR, as Assessed Using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: The CBR was defined as the percentage of participants with a confirmed CR, PR, or SD lasting for at least 6 months. CR: Disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalisation of tumour marker level. All lymph nodes must be non-pathological in size (<10 mm short axis). PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: 6 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2, Cohort 1: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 2: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 3: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 4: Entinostat 5 mg Weekly + Pembrolizumab
Number analyzed (Participants) | 18 | 76 | 53 | 37
percentage of participants | 22.2 [6.4 to 47.6] | 14.5 [7.5 to 24.4] | 30.2 [18.3 to 44.3] | 2.7 [0.1 to 14.2]

4. Secondary Outcome: Phase 2: Progression Free Survival (PFS), as Assessed Using irRECIST
Description: PFS was defined as the number of months from randomization to PD or death due to any cause, whichever occurred first. PD: Sum of the diameters (longest for non-nodal lesions, shortest for nodal lesions) of target and new measurable lesions increases ≥20% (compared to nadir), confirmed by a repeat, consecutive observation at least 4 weeks from the date first documented. Number of participants without evidence of progression or death at Month 6 are reported.
Time Frame: 6 months
Population: FAS included all enrolled participants excluding those that did not receive at least 1 dose of entinostat and pembrolizumab or lacked baseline data. Data were censored for PFS analysis based on prespecified analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2, Cohort 1: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 2: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 3: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 4: Entinostat 5 mg Weekly + Pembrolizumab
Number analyzed (Participants) | 18 | 76 | 53 | 37
Participants | 3 | 17 | 20 | 3

5. Secondary Outcome: Phase 2: PFS, as Assessed Using RECIST 1.1
Description: PFS was defined as the number of months from randomization to PD or death due to any cause, whichever occurred first. PD: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm; the appearance of one or more new lesions; and unequivocal progression of existing non-target lesions. Number of participants without evidence of progression or death at Month 6 are reported.
Time Frame: 6 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2, Cohort 1: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 2: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 3: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 4: Entinostat 5 mg Weekly + Pembrolizumab
Number analyzed (Participants) | 18 | 76 | 53 | 37
Participants | 3 | 17 | 17 | 2

6. Secondary Outcome: Phase 2: PFS Duration, as Determined by the Local Investigator Using irRECIST
Description: PFS was defined as the number of months from randomization to PD or death due to any cause, whichever occurred first. PD: Sum of the diameters (longest for non-nodal lesions, shortest for nodal lesions) of target and new measurable lesions increases ≥20% (compared to nadir), confirmed by a repeat, consecutive observation at least 4 weeks from the date first documented. For purposes of analysis, 1 month was considered to be 30.4375 days.
Time Frame: From date of randomization to PD or death due to any cause (up to 765 days)
Population: FAS included all enrolled participants excluding those that did not receive at least 1 dose of entinostat and pembrolizumab or lacked baseline data.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2, Cohort 1: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 2: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 3: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 4: Entinostat 5 mg Weekly + Pembrolizumab
Number analyzed (Participants) | 18 | 76 | 53 | 37
months | 2.76 [1.18 to 4.07] | 2.83 [1.51 to 4.14] | 4.40 [2.79 to 6.97] | 1.91 [1.38 to 2.79]

7. Secondary Outcome: Phase 2: PFS Duration, as Determined by the Local Investigator Using RECIST 1.1
Description: as for outcome 6
Time Frame: From date of randomization to PD or death due to any cause (up to 765 days)
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2, Cohort 1: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 2: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 3: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 4: Entinostat 5 mg Weekly + Pembrolizumab
Number analyzed (Participants) | 18 | 76 | 53 | 37
months | 2.76 [1.18 to 4.07] | 2.69 [1.48 to 4.07] | 2.96 [1.45 to 6.24] | 1.91 [1.38 to 2.79]

8. Secondary Outcome: Phase 2: Overall Survival
Description: Overall survival was defined as the number of months from randomization to the date of death (due to any cause). For purposes of analysis, 1 month was considered to be 30.4375 days.
Time Frame: From date of randomization to the date of death (up to 765 days)
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2, Cohort 1: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 2: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 3: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 4: Entinostat 5 mg Weekly + Pembrolizumab
Number analyzed (Participants) | 18 | 76 | 53 | 37
months | 25.20 [3.58 to NA] — Due to smaller number of participants with an event, the upper limit of 95% confidence interval (CI) could not be calculated. | 11.73 [7.56 to 13.37] | 12.52 [8.51 to 28.25] | 9.79 [6.11 to 14.36]

9. Secondary Outcome: Phase 2: Duration of Response, as Assessed Using irRECIST
Description: Duration of response was defined as number of months from start date of CR or PR (whichever occurred first) and subsequently confirmed, to the first date that recurrent or progressive disease was documented. CR: Disappearance of all target lesions and any pathological lymph nodes (target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalisation of tumour marker level. All lymph nodes must be non-pathological in size (<10 mm short axis). PR: At least a 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters. PD: At least a 20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, sum must also demonstrate an absolute increase of ≥5 mm; appearance of one or more new lesions; and unequivocal progression of existing non-target lesions. For purposes of analysis, 1 month was considered to be 30.4375 days.
Time Frame: From start date of CR or PR to date of progression (up to 765 days)
Population: FAS included all enrolled participants excluding those that did not receive at least 1 dose of entinostat and pembrolizumab or lacked baseline data. Here, 'Overall number of participants analyzed' = participants who achieved objective response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2, Cohort 1: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 2: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 3: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 4: Entinostat 5 mg Weekly + Pembrolizumab
Number analyzed (Participants) | 4 | 7 | 10 | 2
months | 15.61 [1.18 to NA] — Due to smaller number of participants with an event, the upper limit of 95% CI could not be calculated. | 10.10 [3.94 to NA] — Due to smaller number of participants with an event, the upper limit of 95% CI could not be calculated. | 25.49 [4.60 to 25.49] | 7.33 [NA to NA] — Due to smaller number of participants with an event, the upper and lower limit of 95% CI could not be calculated.

10. Secondary Outcome: Phase 2: Duration of Response, as Assessed Using RECIST 1.1
Description: as for outcome 9
Time Frame: From start date of CR or PR to date of progression (up to 765 days)
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2, Cohort 1: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 2: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 3: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 4: Entinostat 5 mg Weekly + Pembrolizumab
Number analyzed (Participants) | 2 | 7 | 8 | 0
months | NA [NA to NA] — Due to smaller number of participants with an event, median and upper and lower limit of 95% CI could not be calculated. | 10.14 [3.94 to NA] — Due to smaller number of participants with an event, the upper limit of 95% CI could not be calculated. | 25.49 [NA to NA] — Due to smaller number of participants with an event, the upper and lower limit of 95% CI could not be calculated. |

11. Secondary Outcome: Phase 2: Time to Response, as Assessed Using irRECIST
Description: Time to response was defined as the number of months from the randomization date to the first date the participant achieved a PR or CR (whichever response occurred first and was subsequently confirmed). CR: Disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalisation of tumour marker level. All lymph nodes must be non-pathological in size (<10 mm short axis). PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. For purposes of analysis, 1 month was considered to be 30.4375 days.
Time Frame: From the date of randomization to date of PR or CR (up to 765 days)
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2, Cohort 1: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 2: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 3: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 4: Entinostat 5 mg Weekly + Pembrolizumab
Number analyzed (Participants) | 4 | 7 | 10 | 2
months | 4.30 [2.69 to 9.63] | 2.83 [2.69 to 5.49] | 1.95 [1.18 to 2.79] | 4.17 [2.79 to 5.55]

12. Secondary Outcome: Phase 2: Time to Response, as Assessed Using RECIST 1.1
Description: as for outcome 11
Time Frame: From the date of randomization to date of PR or CR (up to 765 days)
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2, Cohort 1: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 2: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 3: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 4: Entinostat 5 mg Weekly + Pembrolizumab
Number analyzed (Participants) | 2 | 7 | 8 | 0
months | 4.29 [2.69 to 5.88] | 2.83 [2.69 to 5.49] | 1.95 [1.18 to 2.79] |

13. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), AEs Resulting in the Permanent Discontinuation of Study Drug, and Death
Description: An adverse event (AE) was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. SAEs included death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized the participant and required medical intervention to prevent 1 of the outcomes listed in this definition. TEAEs were defined as AEs that started on or after the first administration of study drug and within 30 days of the last administration of any study treatment. A summary of serious and non-serious AEs regardless of causality is located in 'Reported Adverse Events module'. For purposes of analysis, 1 month was considered to be 30.4375 days.
Time Frame: From first dose of study drug up to 765 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b (Dose Escalation): Entinostat 3 mg Weekly + Pembrolizumab | Phase 1b (Dose Escalation): Entinostat 5 mg Weekly + Pembrolizumab | Phase 1b (Dose Confirmation): Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 1: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 2: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 3: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 4: Entinostat 5 mg Weekly + Pembrolizumab
Number analyzed (Participants) | 6 | 7 | 9 | 18 | 76 | 53 | 38
Participants
  TEAEs | 6 | 7 | 9 | 18 | 75 | 53 | 37
  SAEs | 4 | 4 | 2 | 10 | 33 | 24 | 14
  AEs Resulting in the Permanent Discontinuation of Study Drug | 1 | 2 | 1 | 7 | 19 | 8 | 7
  AEs Resulting in Death | 1 | 0 | 1 | 3 | 3 | 2 | 1

14. Secondary Outcome: Phase 1b: Number of Participants With at Least One Dose Limiting Toxicities (DLTs)
Description: A DLT was defined as the occurrence of any protocol-specified event in the first cycle of treatment (Day 1 through Day 21) of entinostat in combination with avelumab that were considered by the investigator to be at least possibly related to study drug.
Time Frame: Day 1 through Day 21 (Cycle 1)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b (Dose Escalation): Entinostat 3 mg Weekly + Pembrolizumab | Phase 1b (Dose Escalation): Entinostat 5 mg Weekly + Pembrolizumab | Phase 1b (Dose Confirmation): Entinostat 5 mg Weekly + Pembrolizumab
Number analyzed (Participants) | 6 | 7 | 9
Participants | 0 | 1 | 0

15. Secondary Outcome: Phase 1b: Recommended Phase 2 Dose (RP2D)
Description: The RP2D was determined in discussion with the Sponsor, Medical Monitor, and Dose Determination Phase Investigators. Additionally, observations related to immune correlates, and any cumulative toxicity observed after multiple cycles might be included in the rationale supporting the RP2D. The RP2D could be equal to or less than the preliminary maximum tolerated dose (MTD). The MTD was defined as the highest dose level at which <33% of 6 participants experienced DLT.
Time Frame: Day 1 through Day 21 (Cycle 1)
Population: as for baseline characteristics
Measure: Number; unit: mg
Groups:
- Phase 1b: Entinostat 3 mg or 5 mg Weekly + Pembrolizumab: Participants with NSCLC received entinostat 3 mg or 5 mg administered orally weekly (Days 1, 8, and 15 of each 21-day cycle) along with pembrolizumab 200 mg via IV infusion once every 3 weeks (Day 1 of each 21-day cycle).
Arm/Group | Phase 1b: Entinostat 3 mg or 5 mg Weekly + Pembrolizumab
Number analyzed (Participants) | 22
mg | 5

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 765 days
Description: Safety analysis set included all participants who received at least 1 dose of either study drug, entinostat, or pembrolizumab.
Groups:
- Phase 2, Cohort 3: Entinostat 5 mg Weekly + Pembrolizumab: Participants with melanoma who had previously been treated with and unequivocally progressed on either a PD-1- or PD-L1-blocking antibody, received entinostat 5 mg administered orally weekly (Days 1, 8, and 15 of each 21-day cycle) along with pembrolizumab 200 mgvia IV infusion once every 3 weeks (Day 1 of each 21-day cycle).
Arm/Group | Phase 1b (Dose Escalation): Entinostat 3 mg Weekly + Pembrolizumab | Phase 1b (Dose Escalation): Entinostat 5 mg Weekly + Pembrolizumab | Phase 1b (Dose Confirmation): Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 1: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 2: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 3: Entinostat 5 mg Weekly + Pembrolizumab | Phase 2, Cohort 4: Entinostat 5 mg Weekly + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 6/6 | 0/7 | 1/9 | 8/18 | 41/76 | 31/53 | 25/38
Serious Adverse Events (participants affected / at risk) | 4/6 | 4/7 | 2/9 | 10/18 | 33/76 | 24/53 | 14/38
Other Adverse Events (participants affected / at risk) | 6/6 | 7/7 | 9/9 | 18/18 | 75/76 | 52/53 | 37/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b (Dose Escalation): Entinostat 3 mg Weekly + Pembrolizumab (N=6) | Phase 1b (Dose Escalation): Entinostat 5 mg Weekly + Pembrolizumab (N=7) | Phase 1b (Dose Confirmation): Entinostat 5 mg Weekly + Pembrolizumab (N=9) | Phase 2, Cohort 1: Entinostat 5 mg Weekly + Pembrolizumab (N=18) | Phase 2, Cohort 2: Entinostat 5 mg Weekly + Pembrolizumab (N=76) | Phase 2, Cohort 3: Entinostat 5 mg Weekly + Pembrolizumab (N=53) | Phase 2, Cohort 4: Entinostat 5 mg Weekly + Pembrolizumab (N=38)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 4 | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 3 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1 | 4 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Abdominal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthritis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Encephalitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sialoadenitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 3 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 1 | 1 | 2 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 3 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Death (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Brain mass (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0
Steatohepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spinal cord injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Embolism (Vascular disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hypercalcaemia of malignancy (Endocrine disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b (Dose Escalation): Entinostat 3 mg Weekly + Pembrolizumab (N=6) | Phase 1b (Dose Escalation): Entinostat 5 mg Weekly + Pembrolizumab (N=7) | Phase 1b (Dose Confirmation): Entinostat 5 mg Weekly + Pembrolizumab (N=9) | Phase 2, Cohort 1: Entinostat 5 mg Weekly + Pembrolizumab (N=18) | Phase 2, Cohort 2: Entinostat 5 mg Weekly + Pembrolizumab (N=76) | Phase 2, Cohort 3: Entinostat 5 mg Weekly + Pembrolizumab (N=53) | Phase 2, Cohort 4: Entinostat 5 mg Weekly + Pembrolizumab (N=38)
Fatigue (General disorders) | 2 | 6 | 6 | 14 | 36 | 29 | 22
Oedema peripheral (General disorders) | 1 | 1 | 0 | 3 | 10 | 10 | 2
Pyrexia (General disorders) | 2 | 0 | 1 | 3 | 9 | 9 | 1
Pain (General disorders) | 1 | 2 | 2 | 3 | 10 | 4 | 1
Chills (General disorders) | 0 | 0 | 1 | 1 | 3 | 7 | 4
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 1 | 4 | 5 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 5 | 5 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 2 | 4 | 1 | 2
Oedema (General disorders) | 0 | 0 | 0 | 1 | 4 | 3 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 3
Malaise (General disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 2
Mucosal inflammation (General disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 3
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Nodule (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Tenderness (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Early satiety (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Induration (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infusion site bruising (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Temperature intolerance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 1 | 3 | 5 | 21 | 30 | 9
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 3 | 5 | 25 | 20 | 13
Vomiting (Gastrointestinal disorders) | 2 | 0 | 3 | 4 | 15 | 13 | 8
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 13 | 16 | 9
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 8 | 8 | 11
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 8 | 3 | 5
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 3 | 1 | 5 | 3 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 3 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 3
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 3 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 2
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oesophageal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Reactive gastropathy (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0 | 5 | 3 | 27 | 16 | 10
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 4 | 20 | 14 | 7
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 14 | 10 | 8
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 5 | 19 | 4 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 5 | 11 | 7 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 7 | 3 | 5
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 4 | 9 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 4 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 5 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 2 | 2 | 2
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 3 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 2 | 2 | 20 | 8 | 10
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 2 | 15 | 8 | 14
Platelet count decreased (Investigations) | 0 | 1 | 0 | 4 | 12 | 9 | 8
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 2 | 9 | 9 | 9
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 7 | 7 | 9
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 2 | 2 | 10 | 3
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 1 | 4 | 9 | 3
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 5 | 5 | 5
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 4 | 4 | 3
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 5 | 2 | 2
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 4 | 2
Weight increased (Investigations) | 0 | 1 | 0 | 1 | 1 | 1 | 1
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Electrocardiogram QT interval (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Antineutrophil cytoplasmic antibody decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood alkaline phosphatase (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Carbon dioxide increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Differential white blood cell count abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eosinophil count increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Glucose urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intraocular pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Platelet count (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Protein total decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thyroxine free increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tri-iodothyronine decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 3 | 17 | 21 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 3 | 7 | 15 | 10 | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 3 | 4 | 2 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2 | 4 | 2 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2 | 4 | 2 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 6 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 3 | 3 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 4 | 0 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2 | 2 | 2
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal and connective tissue disorders (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 10 | 34 | 24 | 17
Arthralgia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 5 | 10 | 8 | 9
Back pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 3 | 15 | 8 | 3
Myalgia (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 4 | 4 | 7 | 6
Pain in extremity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 5 | 5 | 3
Muscular weakness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 5 | 5 | 1
Muscle spasms (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 4
Musculoskeletal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 5 | 3 | 0
Neck pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 3 | 2
Groin pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 2
Musculoskeletal chest pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 3 | 1 | 0
Flank pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 3
Joint swelling (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Bone pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Muscle atrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Pain in jaw (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0
Limb discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle twitching (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal stiffness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myopathy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myositis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neck mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Osteonecrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Soft tissue disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Spinal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 3 | 22 | 13 | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 6 | 5 | 3
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 1 | 5 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 3 | 6 | 13 | 7
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1 | 9 | 12 | 6
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 2 | 6 | 4
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 2 | 3 | 3
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 2 | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myasthenia gravis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Orthostatic intolerance (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Paraplegia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Visual field defect (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vocal cord paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3 | 1 | 4 | 6 | 12 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2 | 2 | 8 | 4
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 4 | 7 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 3 | 3 | 1 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0 | 5 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 3 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 5 | 2 | 3
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 4 | 2 | 2
Lung infection (Infections and infestations) | 0 | 1 | 0 | 3 | 4 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 5 | 1
Oral candidiasis (Infections and infestations) | 0 | 1 | 1 | 3 | 3 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 2 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 4 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 2 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fungal oesophagitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Groin abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mastoiditis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tinea cruris (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tinea infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 1 | 2 | 5 | 8 | 5
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 6
Depression (Psychiatric disorders) | 0 | 1 | 0 | 2 | 2 | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 8 | 4 | 3
Embolism (Vascular disorders) | 1 | 0 | 0 | 0 | 2 | 2 | 1
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Penetrating atherosclerotic ulcer (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Poor venous access (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 3 | 5 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 5 | 2 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 2 | 4 | 1 | 2
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 4 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bundle branch block left (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 5 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 2 | 2
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 3 | 2 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye disorder (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eyelid function disorder (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eyelid ptosis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 1 | 3 | 2 | 3
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 3
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Inner ear disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Perineal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vaginal lesion (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Allergy to arthropod sting (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Autoimmune disorder (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Steatohepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infection prophylaxis (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus operation (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wound drainage (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of the results of the multi-center Study shall not be made before the first multi-site publication by Sponsor or Publications Committee. No Public Presentation by Institution or Investigator will be made until Study Documentation/Results from all sites are received and analyzed by Sponsor. Separate publication by Investigator will be delayed for a period of 18 months until the initial publication by Committee or Sponsor, or a determination is made not to make such publication.

DOCUMENTS (2):
  • Study Protocol (2018-04-12): https://cdn.clinicaltrials.gov/large-docs/36/NCT02437136/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-26): https://cdn.clinicaltrials.gov/large-docs/36/NCT02437136/SAP_001.pdf